CLINICAL TRIAL: NCT05184309
Title: Effects of Serious Games for Shoulder Rehabilitation and Measurement of Approximation Force: Randomized Controlled Trial
Brief Title: Effects of Serious Games for Shoulder Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medipolftr
Record Dates: First submitted 2021-12-26; First posted 2022-01-11 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Serious Game; Rotator Cuff Tears; Rehabilitation
Keywords: Serious game; Rotator cuff rupture; Shoulder Rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded in enrollment and assessment process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercise group (Experimental): Conventional Exercises
  Interventions: Other: ConventioanalExercises
- Serious game group (Experimental): Serious Games
  Interventions: Other: Serious games

INTERVENTIONS:
Other: ConventioanalExercises — Wand exercises and shoulder wheel exercises to increase the range of motion of the shoulder joint with 10 repetitions will be applied in CEG. Finger ladder exercises will be performed in the abduction and flexion position with 5 repetitions, holding the endpoint for 5 seconds. Stretching exercises with 5 repetitions will be applied in all directions for the limitation of movement, holding it for 20 seconds at the endpoint. Individuals performed conventional exercises twice a week for 6 weeks.
  Arms: Conventional exercise group
Other: Serious games — A Serious game program will be applied to the individuals twice a week for 6 weeks in this group. Armrotate, Uball, Balance Surf and Balance Adventure games will be developed by Becure company for shoulder rehabilitation. These games developed for shoulder rehabilitation will be applied to individuals under the supervision of a physiotherapist. Each game will be played for 10 minutes, for a total of 40 minutes.
  Arms: Serious game group

SUMMARY:
The aim of this study is to examine the effect of Serious-Game Exercise (SGE) platform on pain, range of motion (ROM), joint position sense, shoulder functions, and approximation force in patients with rotator cuff rupture. In addition, another objective is to evaluate the usage of balance board as a measurement tool for measuring the approximation force in the rotator cuff rupture.

DETAILED DESCRIPTION:
Purpose: To examine the effect of Serious-Game Exercise (SGE) platform on pain, range of motion (ROM), joint position sense, shoulder functions, and approximation force in patients with rotator cuff rupture. In addition, another objective is to evaluate the usage of balance board as a measurement tool for measuring the approximation force in the rotator cuff rupture.

Method: Twenty patients with rotator cuff rupture will be included in the study. They will be divided into two groups as a serious game group (SGG) and a conventional exercise group (CEG) with a randomization method. The Serious game exercise program developed for shoulder rehabilitation will be applied to the SG group and conventional exercise training will be applied to the CEG. Pain severity, flexion, abduction and external rotation ROM, functionality, joint position sense, and approximation force of all individuals will be evaluated pre and post-treatment. SGG and CEG underwent serious games and conventional therapy twice a week for 6 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 40-60,
* having pain for more than 4 weeks,
* not having had any shoulder surgery

Exclusion Criteria:

* Individuals with cervical-origin neurological findings, uncooperative, different orthopedic problems in the same shoulder,
* neurological, vascular and cardiac problems that limit function

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment- Visual Analogue scale | 5 minutes
  Pain level is measured with the visual analogue scale (VAS), at rest and activity. The visual analogue scale consists of a 10-cm line. Participants were asked to indicate in the scale their current level of pain where the higher values are more intense pain.
Range of motion | 5 minutes
  The range of motion of the joint of the individuals participating in the study will be evaluated with Becure Extremity ROM. The patient stands in front of the camera and perform the directed movement. In this study, flexion, abduction and external rotation ranges of motion of the shoulder joint will be measured.
Joint position sense | 5 minutes
  The joint position sense of the individuals will be evaluated with the Becure Extremity ROM. Subjects will be first asked to raise their shoulder to a certain degree and bring it to the same angle value with eyes closed. The difference between shoulder angles will be calculated by recording the angle value formed with eyes closed and open.
Shoulder approximation force | 5 minutes
  Shoulder approximation force will be evaluated with the Becure Balance System. During this measurement, the individual will be asked to put both hands on the Balance Board and then apply downward force without using body weight. Measurements will be taken in standing and sitting positions (0° and 90°).

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | 5 minutes
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used to evaluate the limitations and functionality of the individuals with upper extremity problems. The DASH that includes 30 questions and 3 sections is used to evaluate symptoms, parameters such as social function, work, sleep and self-confidence of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
When the study will be published in a journal, all of researchers can see the result of the participants of this study.

REFERENCES:
- [Result] Pekyavas NO, Ergun N. Comparison of virtual reality exergaming and home exercise programs in patients with subacromial impingement syndrome and scapular dyskinesis: Short term effect. Acta Orthop Traumatol Turc. 2017 May;51(3):238-242. doi: 10.1016/j.aott.2017.03.008. Epub 2017 Apr 24. PMID 28446376
- See also: Comparison of virtual reality exergaming and home exercise programs in patients with subacromial impingement syndrome and scapular dyskinesis: Short term effect — https://pubmed.ncbi.nlm.nih.gov/28446376/
- Available data/document: Statistical Analysis Plan: Principle investigator — https://pubmed.ncbi.nlm.nih.gov/28446376/